CLINICAL TRIAL: NCT02096055
Title: Four-Arm Randomized Phase II Study of SGI-110: 5 Days, Versus 10 Days, Versus 5 Days + Idarubicin, Versus 5 Days + Cladribine, in Previously Untreated Patients >/= 70 Years With Acute Myeloid Leukemia
Brief Title: Guadecitabine With or Without Idarubicin or Cladribine in Treating Older Patients With Previously Untreated Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0843; NCI-2014-00981 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2013-0843 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2014-03-20; First posted 2014-03-26 (Estimated); Results first posted 2022-05-24 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Untreated Adult Acute Myeloid Leukemia
MeSH Terms: interventions — Cladribine; guadecitabine; Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm I (guadecitabine) (Experimental): INDUCTION THERAPY: Patients receive guadecitabine SC on days 1-5. Courses repeat every 4-6 weeks for 2-3 courses in the absence of disease progression or unacceptable toxicity. Patients achieving a CR or CRp continue on to Maintenance therapy; patients not achieving CR or CRi but deriving clinical benefit may continue to Maintenance therapy at the discretion of the PI.
  MAINTENANCE THERAPY: Patients receive guadecitabine as in Induction therapy. Courses repeat every 4-8 weeks for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Guadecitabine
- Arm II (CLOSED) (guadecitabine) (Experimental): INDUCTION THERAPY: Patients receive guadecitabine SC on days 1-10. Courses repeat every 4-6 weeks for 2-3 courses in the absence of disease progression or unacceptable toxicity. Patients achieving a CR or CRp continue on to Maintenance therapy; patients not achieving CR or CRi but deriving clinical benefit may continue to Maintenance therapy at the discretion of the PI.
  MAINTENANCE THERAPY: Patients receive guadecitabine SC on days 1-5 (days 1-10 of courses 1 and 2). Courses repeat every 4-8 weeks for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Guadecitabine
- Arm III (guadecitabine, idarubicin) (Experimental): INDUCTION THERAPY: Patients receive guadecitabine SC on days 1-5 and idarubicin IV over up to 1 hour on days 1-2. Courses repeat every 4-6 weeks for 2-3 courses in the absence of disease progression or unacceptable toxicity. Patients achieving a CR or CRp continue on to Maintenance therapy; patients not achieving CR or CRi but deriving clinical benefit may continue to Maintenance therapy at the discretion of the PI.
  MAINTENANCE THERAPY: Patients receive guadecitabine SC on days 1-5 and idarubicin IV over up to 1 hour on day 1. Courses repeat every 4-8 weeks for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Guadecitabine; Drug: Idarubicin
- Arm IV (CLOSED) (guadecitabine, cladribine) (Experimental): INDUCTION THERPAY: Patients receive guadecitabine SC and cladribine IV over up to 1 hour on days 1-5. Courses repeat every 4-6 weeks for 2-3 courses in the absence of disease progression or unacceptable toxicity. Patients achieving a CR or CRp continue on to Maintenance therapy; patients not achieving CR or CRi but deriving clinical benefit may continue to Maintenance therapy at the discretion of the PI.
  MAINTENANCE THERAPY: Patients receive guadecitabine SC and cladribine IV over up to 1 hour on days 1-5. Courses repeat every 4-8 weeks for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cladribine; Drug: Guadecitabine

INTERVENTIONS:
Drug: Cladribine — Given IV
  Other Names: 2-CdA; 2CDA; CdA; Cladribina; Leustat; Leustatin; Leustatine; RWJ-26251
  Arms: Arm IV (CLOSED) (guadecitabine, cladribine)
Drug: Guadecitabine — Given SC
  Other Names: DNMT inhibitor SGI-110; S110; SGI-110
Drug: Idarubicin — Given IV
  Other Names: 4-Demethoxydaunomycin; 4-demethoxydaunorubicin; 4-DMDR
  Arms: Arm III (guadecitabine, idarubicin)

SUMMARY:
This randomized phase II trial studies how well guadecitabine with or without idarubicin or cladribine works in treating older patients with previously untreated acute myeloid leukemia. Guadecitabine may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as idarubicin and cladribine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether guadecitabine with or without idarubicin or cladribine is more effective in treating older patients with previously untreated acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the complete remission (CR) rate, remission duration, leukemia-free survival, and survival in patients >= 70 years with previously untreated acute myeloid leukemia (AML) with 4 different guadecitabine (SGI-110) single agent and SGI-110 based combination regimens.

II. To determine the safety profile and tolerability of the 4 SGI-110 single agent and SGI-110 based combination regimens in patients >= 70 years of age with previously untreated AML.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I:

INDUCTION THERAPY: Patients receive guadecitabine subcutaneously (SC) on days 1-5. Courses repeat every 4-6 weeks for 2-3 courses in the absence of disease progression or unacceptable toxicity. Patients achieving a CR or CR with incomplete platelet recovery (CRp) continue on to Maintenance therapy; patients not achieving CR or complete remission with incomplete hematologic recovery (CRi) but deriving clinical benefit may continue to Maintenance therapy at the discretion of the Principal Investigator (PI).

MAINTENANCE THERAPY: Patients receive guadecitabine as in Induction therapy. Courses repeat every 4-8 weeks for up to 24 months in the absence of disease progression or unacceptable toxicity.

ARM II (CLOSED):

INDUCTION THERAPY: Patients receive guadecitabine SC on days 1-10. Courses repeat every 4-6 weeks for 2-3 courses in the absence of disease progression or unacceptable toxicity. Patients achieving a CR or CRp continue on to Maintenance therapy; patients not achieving CR or CRi but deriving clinical benefit may continue to Maintenance therapy at the discretion of the PI.

MAINTENANCE THERAPY: Patients receive guadecitabine SC on days 1-5 (days 1-10 of courses 1 and 2). Courses repeat every 4-8 weeks for up to 24 months in the absence of disease progression or unacceptable toxicity.

ARM III:

INDUCTION THERAPY: Patients receive guadecitabine SC on days 1-5 and idarubicin intravenously (IV) over up to 1 hour on days 1-2. Courses repeat every 4-6 weeks for 2-3 courses in the absence of disease progression or unacceptable toxicity. Patients achieving a CR or CRp continue on to Maintenance therapy; patients not achieving CR or CRi but deriving clinical benefit may continue to Maintenance therapy at the discretion of the PI.

MAINTENANCE THERAPY: Patients receive guadecitabine SC on days 1-5 and idarubicin IV over up to 1 hour on day 1. Courses repeat every 4-8 weeks for up to 24 months in the absence of disease progression or unacceptable toxicity.

ARM IV (CLOSED):

INDUCTION THERAPY: Patients receive guadecitabine SC and cladribine IV over up to 1 hour on days 1-5. Courses repeat every 4-6 weeks for 2-3 courses in the absence of disease progression or unacceptable toxicity. Patients achieving a CR or CRp continue on to Maintenance therapy; patients not achieving CR or CRi but deriving clinical benefit may continue to Maintenance therapy at the discretion of the PI.

MAINTENANCE THERAPY: Patients receive guadecitabine SC and cladribine IV over up to 1 hour on days 1-5. Courses repeat every 4-8 weeks for up to 24 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every month.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated AML patients, except those who have received prior therapy with hydroxyurea, single agent chemotherapy (e.g. decitabine), hematopoietic growth factors, biological or targeted therapies are allowed
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Sign a written informed consent form
* Total bilirubin =< 2 mg/dL
* Serum glutamate pyruvate transaminase (SGPT) or serum glutamic oxaloacetic transaminase (SGOT) =< 4 x upper limit of normal (ULN)
* Creatinine clearance of >= 50 mL/min (estimated by the Cockcroft-Gault [C-G] formula)
* Male patients must use an effective contraceptive method during the study and for a minimum of 8 weeks after study treatment
* Baseline left ventricular ejection fraction (LVEF) >= 40%

Exclusion Criteria:

* Patients with >= New York Heart Association (NYHA) grade 3 heart disease as assessed by history and/or physical examination
* Patients who received more than one full course of prior hypomethylating agents azacitidine or decitabine
* Have any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver, or other organ system that may place the patient at undue risk to undergo treatment
* Patients with a systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment)
* Pregnant or lactating patients
* Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results
* Any concurrent malignancy with the exception of the following: a) patients with treated non-melanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia, regardless of the disease-free duration, are eligible for this study if definitive treatment for the condition has been completed; b) patients with organ-confined prostate cancer with no evidence of recurrent or progressive disease based on prostate-specific antigen (PSA) values are also eligible for this study if hormonal therapy has been initiated or a radical prostatectomy has been performed

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-04-04 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2020-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hagop M Kantarjian, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: April 2014 to July 2018
Groups:
- Arm I (Guadecitabine) x 5 Days: INDUCTION THERAPY: Patients receive guadecitabine SC on days 1-5. Courses repeat every 4-6 weeks for 2-3 courses in the absence of disease progression or unacceptable toxicity. Patients achieving a CR or CRp continue on to Maintenance therapy; patients not achieving CR or CRi but deriving clinical benefit may continue to Maintenance therapy at the discretion of the PI.
  MAINTENANCE THERAPY: Patients receive guadecitabine as in Induction therapy. Courses repeat every 4-8 weeks for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Guadecitabine: Given SC
- Arm II (CLOSED) (Guadecitabine) x 10 Days: INDUCTION THERAPY: Patients receive guadecitabine SC on days 1-10. Courses repeat every 4-6 weeks for 2-3 courses in the absence of disease progression or unacceptable toxicity. Patients achieving a CR or CRp continue on to Maintenance therapy; patients not achieving CR or CRi but deriving clinical benefit may continue to Maintenance therapy at the discretion of the PI.
  MAINTENANCE THERAPY: Patients receive guadecitabine SC on days 1-5 (days 1-10 of courses 1 and 2). Courses repeat every 4-8 weeks for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Guadecitabine: Given SC
- Arm III (Guadecitabine, Idarubicin): INDUCTION THERAPY: Patients receive guadecitabine SC on days 1-5 and idarubicin IV over up to 1 hour on days 1-2. Courses repeat every 4-6 weeks for 2-3 courses in the absence of disease progression or unacceptable toxicity. Patients achieving a CR or CRp continue on to Maintenance therapy; patients not achieving CR or CRi but deriving clinical benefit may continue to Maintenance therapy at the discretion of the PI.
  MAINTENANCE THERAPY: Patients receive guadecitabine SC on days 1-5 and idarubicin IV over up to 1 hour on day 1. Courses repeat every 4-8 weeks for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Guadecitabine: Given SC
  Idarubicin: Given IV
- Arm IV (CLOSED) (Guadecitabine, Cladribine): INDUCTION THERPAY: Patients receive guadecitabine SC and cladribine IV over up to 1 hour on days 1-5. Courses repeat every 4-6 weeks for 2-3 courses in the absence of disease progression or unacceptable toxicity. Patients achieving a CR or CRp continue on to Maintenance therapy; patients not achieving CR or CRi but deriving clinical benefit may continue to Maintenance therapy at the discretion of the PI.
  MAINTENANCE THERAPY: Patients receive guadecitabine SC and cladribine IV over up to 1 hour on days 1-5. Courses repeat every 4-8 weeks for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Cladribine: Given IV
  Guadecitabine: Given SC
Period: Overall Study
Arm/Group | Arm I (Guadecitabine) x 5 Days | Arm II (CLOSED) (Guadecitabine) x 10 Days | Arm III (Guadecitabine, Idarubicin) | Arm IV (CLOSED) (Guadecitabine, Cladribine)
Started | 13 | 9 | 13 | 9
Completed | 13 | 9 | 13 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Guadecitabine) x 5 Days | Arm II (CLOSED) (Guadecitabine) x 10 Days | Arm III (Guadecitabine, Idarubicin) | Arm IV (CLOSED) (Guadecitabine, Cladribine) | Total
Number analyzed (Participants) | 13 | 9 | 13 | 9 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 13 | 9 | 13 | 9 | 44
Age, Continuous [Median (Full Range); unit: years] | 73 [70 to 81] | 76 [71 to 83] | 75 [71 to 82] | 76 [70 to 82] | 75 [70 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 4 | 2 | 12
  Male | 11 | 5 | 9 | 7 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 11 | 8 | 13 | 9 | 41
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 13 | 9 | 13 | 9 | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Complete Response
Description: Complete Response = Complete Remission (CR) + Complete Remission without blood count recovery (CRi) - CR: Neutrophil count >/= 1.0 x 10^9/L and platelet count >/= 100 x 10^9/L, and normal bone marrow differential (</+ 5% blasts). (CRi): Peripheral blood and bonemarrow results as for CR, but with platelet counts of < 100 x 109/L or ANC < 1.0 x 109/L
Time Frame: Up to 4 years, 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Guadecitabine) x 5 Days | Arm II (CLOSED) (Guadecitabine) x 10 Days | Arm III (Guadecitabine, Idarubicin) | Arm IV (CLOSED) (Guadecitabine, Cladribine)
Number analyzed (Participants) | 13 | 9 | 13 | 9
Participants | 5 | 5 | 10 | 0

2. Primary Outcome: Remission Duration
Description: The date of Complete Response to the date of loss of response or last follow-up.
Time Frame: Up to 4 years, 3 months
Population: Zero participants in the guadecitabine + Cladribine arm had a Complete Response.
Measure: Median (Full Range); unit: Months
Arm/Group | Arm I (Guadecitabine) x 5 Days | Arm II (CLOSED) (Guadecitabine) x 10 Days | Arm III (Guadecitabine, Idarubicin) | Arm IV (CLOSED) (Guadecitabine, Cladribine)
Number analyzed (Participants) | 5 | 5 | 10 | 0
Months | 7.4 [1.2 to 12.6] | 14.2 [5.7 to 19.0] | 5.3 [1.4 to 37.0] |

3. Primary Outcome: Leukemia-free Survival
Description: Survival time will be estimated using the Kaplan-Meier method. The two-sided log-rank test will be used to assess the differences of time to events between groups. Time from date of treatment start until the date of first objective documentation of disease-relapse.
Time Frame: Up to 4 years, 3 months
Measure: Median (Full Range); unit: Months
Arm/Group | Arm I (Guadecitabine) x 5 Days | Arm II (CLOSED) (Guadecitabine) x 10 Days | Arm III (Guadecitabine, Idarubicin) | Arm IV (CLOSED) (Guadecitabine, Cladribine)
Number analyzed (Participants) | 13 | 9 | 13 | 9
Months | 4.2 [2.1 to 13.9] | 10.0 [0.5 to 21.7] | 7.4 [2.0 to 39.5] | 4.3 [1.1 to 28.9]

4. Primary Outcome: Survival
Description: Survival time will be estimated using the Kaplan-Meier method. The two-sided log-rank test will be used to assess the differences of time to events between groups.
Time Frame: Up to 4 years, 3 months
Measure: Median (Full Range); unit: Months
Arm/Group | Arm I (Guadecitabine) x 5 Days | Arm II (CLOSED) (Guadecitabine) x 10 Days | Arm III (Guadecitabine, Idarubicin) | Arm IV (CLOSED) (Guadecitabine, Cladribine)
Number analyzed (Participants) | 13 | 9 | 13 | 9
Months | 13.1 [3.3 to 28.8] | 13.0 [0.5 to 43.8] | 15.4 [2.0 to 47.0] | 11.9 [1.9 to 28.9]

5. Primary Outcome: Number of Participants With the Most Frequently Reports Grade 3 or 4 Adverse Event.
Description: The most frequently reported adverse events will be determined by the Principal Investigator. The number of participants who experienced the most frequent grade 3 or 4 adverse events will be reported.
Time Frame: Up to 4 years, 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Guadecitabine) x 5 Days | Arm II (CLOSED) (Guadecitabine) x 10 Days | Arm III (Guadecitabine, Idarubicin) | Arm IV (CLOSED) (Guadecitabine, Cladribine)
Number analyzed (Participants) | 13 | 9 | 13 | 9
Participants
  Infection/Sepsis | 4 | 8 | 8 | 9
  Febrile Neutropenia | 5 | 2 | 4 | 9
  Fatigue | 0 | 0 | 3 | 0

ADVERSE EVENTS:
Time Frame: Up to 4 years, 3 months
Arm/Group | Arm I (Guadecitabine) x 5 Days | Arm II (CLOSED) (Guadecitabine) x 10 Days | Arm III (Guadecitabine, Idarubicin) | Arm IV (CLOSED) (Guadecitabine, Cladribine)
All-Cause Mortality (participants affected / at risk) | 2/13 | 1/9 | 1/13 | 2/9
Serious Adverse Events (participants affected / at risk) | 9/13 | 7/9 | 10/13 | 6/9
Other Adverse Events (participants affected / at risk) | 13/13 | 7/9 | 13/13 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Guadecitabine) x 5 Days (N=13) | Arm II (CLOSED) (Guadecitabine) x 10 Days (N=9) | Arm III (Guadecitabine, Idarubicin) (N=13) | Arm IV (CLOSED) (Guadecitabine, Cladribine) (N=9)
Acute Coronary Syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back Pain (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Breast Infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Bronchopulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenic Fever (Blood and lymphatic system disorders) | 4 (7) | 2 (3) | 4 (5) | 6 (9)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gallbladder infection (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart Failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 4 (4) | 3 (3) | 3 (3) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pain Extremity (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic Event (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infeciton (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Guadecitabine) x 5 Days (N=13) | Arm II (CLOSED) (Guadecitabine) x 10 Days (N=9) | Arm III (Guadecitabine, Idarubicin) (N=13) | Arm IV (CLOSED) (Guadecitabine, Cladribine) (N=9)
Allergy (Immune system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bladder Spasms (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac Ischemia/Infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 6 (6) | 4 (4)
Constitutional Symptoms (General disorders) | 2 (2) | 3 (4) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dermatology Skin/Other (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 6 (6) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema Limb (General disorders) | 3 (3) | 4 (4) | 7 (7) | 1 (1)
Elevated Alanine Aminotransferase (Investigations) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Elevated Aspartate Aminotransferase (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (1) | 4 (4) | 2 (2)
Fever (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flu-like syndrome (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage (General disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Hyperbillirubinemia (Investigations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 3 (5) | 7 (14) | 8 (15) | 6 (11)
Insomnia (Psychiatric disorders) | 4 (4) | 0 (0) | 4 (4) | 0 (0)
Memory Impairment (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (5)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal/Soft Tissue-Other (Specify) (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Myositis (inflammation/damage of muscle) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (3) | 5 (5)
Neurology-Other (Specify) (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Neutropenia (Investigations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Neutropenic Fever (Blood and lymphatic system disorders) | 4 (6) | 1 (2) | 4 (4) | 7 (10)
Obstruction GI (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 2 (2) | 2 (2) | 4 (6) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1) | 2 (2) | 2 (2)
Rash: dermatitis associated with radiation--Select (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sweating (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
thrombocytopenia (Investigations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1 (1) | 2 (3) | 4 (4) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular arrhythmia--Select (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Weight Loss (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-03): https://cdn.clinicaltrials.gov/large-docs/55/NCT02096055/Prot_SAP_000.pdf